CLINICAL TRIAL: NCT02398058
Title: A Phase Ib Study on the Combination of Trabectedin and Olaparib in Unresectable Advanced/Metastatic Sarcomas After Failure of Standard Therapies
Brief Title: Trabectedin Plus Olaparib in Metastatic or Advanced Sarcomas (TOMAS)
Acronym: TOMAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: PharmaMar (Industry); AstraZeneca (Industry); Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOMAS; 2013-003638-33 (EudraCT Number)
Record Dates: First submitted 2015-01-14; First posted 2015-03-25 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Soft Tissue Sarcoma; Bone Tumor
Keywords: trabectedin; olaparib; sarcoma; bone tumor
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Trabectedin; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trabectedin plus olaparib (Experimental): All patients will be treated with trabectedin and olaparib in an open-label fashion.
  The dosage of the drugs at which each patient is treated depends on the dose level reached at the time of enrollment.
  Interventions: Drug: trabectedin; Drug: olaparib

INTERVENTIONS:
Drug: trabectedin — trabectedin will be administered in a 24-h continuous i.v. infusion every 3 weeks
  Other Names: ET-743; Yondelis
Drug: olaparib — olaparib will be administered in a continuous daily dose every 12 hours
  Other Names: AZD-2281; Lynparza

SUMMARY:
This is a Phase 1b, multi-site, open-label, non-randomized clinical trial evaluating the safety, tolerability, and pharmacokinetics of escalating doses of olaparib and trabectedin in patients with unresectable advanced/metastatic sarcomas. Patients will continue to be treated on this combination regimen in the absence of disease progression, intolerable toxicity or patient's decision.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* histologically documented and not surgically resectable or metastatic sarcomas which progressed after first or further line treatments for relapsing disease
* Measurable disease as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0/1. ECOG PS 2 are eligible if depends solely on orthopedic problems
* Estimated life expectancy of ≥ 4 months
* Age ≥18 years
* Adequate organ function: Hemoglobin > 10.0 g/dl; Absolute neutrophil count (ANC) >1,500/mm3; Platelet count >= 100,000/μl; Total bilirubin < 1.5 times the upper limit of normal (ULN); ALT and AST < 2.5 x ULN (< 5 x ULN for patients with liver involvement of their cancer); Alkaline phosphatase < 2.5 x ULN; PT-INR/PTT < 1.5 x ULN; Serum creatinine < 1.5 x ULN or creatinine clearance ≥ 50 ml/min; Albumin > 25 g/l; Creatine phosphokinase (CPK) < 2.5 x ULN

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Previous enrolment in the present study
* Participation in another clinical study with an investigational product during the last month
* Persistent toxicities (≥CTCAE grade 2) with the exception of alopecia, caused by previous anticancer therapies
* Dementia or significantly altered mental status
* Patients with any severe and/or uncontrolled medical conditions
* HIV infection
* Active clinically serious infections (> grade 2 NCI-CTCAE version 4.03).
* Active viral hepatitis (HBV or HCV infection)
* Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, does not require corticosteroid treatment, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry).
* Patients with seizure disorders requiring medication (such as steroids or anti-epileptics)
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days before the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 5 months after last dose of study drug
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Patients unable to swallow oral medications
* Uncontrolled diabetes (fasting glucose > 2 x ULN)
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent (except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg for adrenal insufficiency). Topical or inhaled corticosteroids are permitted
* Patients with a history of another malignancy within 5 years prior to study entry, except curatively treated non-melanotic skin cancer or in-situ cervical cancer or other solid tumors curatively treated with no evidence of disease for ≥5 years.
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of treatment start
* Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy allowed)
* Major surgery within 4 weeks of start of study
* Prior exposure to the study drugs or their analogues
* Patients with known hypersensitivity to trabectedin, olaparib or to their excipients
* Patients can receive a stable dose of bisphosphonates for bone metastases before and during the study as long as these were started at least 4 weeks prior to treatment with the study drugs
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* A history of noncompliance to medical regimens or inability or unwillingness to return for scheduled visits
* Corrected QT interval on the 12-lead ECG (QTc) >470 msec (Bazett Formula)
* use of strong CYP3A4 inhibitors/inducers
* Patients with myelodysplastic syndrome/acute myeloid leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07-20 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | from start up to 6 weeks
  safety will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.03

SECONDARY OUTCOMES:
Best Overall Response | baseline and every 2 cycles (6 weeks +/- 1 week) up to 2 years
  best overall response will be defined according to the Response Evaluation Criteria in Solid Tumor version 1.1 (RECIST v 1.1)
Clinical Benefit Rate | baseline and every 2 cycles (6 weeks +/- 1 week) up to 2 years
  Clinical Benefit Rate (CBR): will be defined as the rate of CR (complete response) + PR (partial response) + stable disease lasting at least 12 weeks. CR, PR and stable disease will be defined according to RECIST v 1.1.
Growth Modulation Index | baseline and every 2 cycles (6 weeks +/- 1 week) up to 2 years
  Growth modulation index (GMI) will be calculated as: GMI=TTPn/TTPn-1. TTPn: Time To Progression on the new agent. TTP n-1: Time To Progression on the treatment the patient received just before the new agent was started.
Overall Survival | baseline and up to 2 years
  time from the date of enrollment to date of death or to the date being censored at two years (whichever occurs first).
Duration of Tumor Response | baseline and every 2 cycles (6 weeks +/- 1 week) up to 2 years
  Duration of Objective Response (complete or partial responses) will be measured from the date that a complete or partial response is first documented (whichever occurs first) to date of progression or death due to progressive disease, whichever occurs first.
Progression-Free Survival (PFS) | baseline and every 2 cycles (6 weeks +/- 1 week) up to 2 years
  PFS is defined as the time from the date of enrollment to the date of first documentation of disease progression, or to the death from any cause.
Pharmacokinetic of trabectedin (AUC) | baseline, days 1-2-3-4-5-8-15 of the first two cycles
  The concentration-time data will be used for a preliminary assessment of the effect of combination therapy on the single-dose pharmacokinetics of trabectedin and olaparib. The data will be analyzed by noncompartmental methods. Pharmacokinetic parameters for trabectedin: steady state profile, end of infusion concentration, area under the concentration-time curve (AUC), and, if data permit, terminal phase half-life. For these parameters, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean. Any drug-drug interaction will be thoroughly searched. For both trabectedin and olaparib all pharmacokinetic evaluations will be done only for the first 2 cycles.
Pharmacokinetic of olaparib (steady state profile and so maximum concentration, minimal concentration, and AUC will be calculated) | baseline, day -5 cycle 1, day 1 cycle 2, of the first two cycles
  The concentration-time data will be used for a preliminary assessment of the effect of combination therapy on the single-dose pharmacokinetics of trabectedin and olaparib. The data will be analyzed by noncompartmental methods. The following pharmacokinetic parameter values will be obtained for olaparib: steady state profile and so maximum concentration, minimal concentration, and AUC will be calculated. For these parameters, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean. Any drug-drug interaction will be thoroughly searched. For both trabectedin and olaparib all pharmacokinetic evaluations will be done only for the first 2 cycles.
safety evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 | baseline up to 28 days after last dose of study treatment up to 2 years
  safety will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.03
Biomarkers (composite outcome) | baseline, day 1-2-8-15 of each cycle up to 2 years
  Several gene assessments (expression, amplification/ deletion, single nucleotide polymorphisms) on DNA-damage response-related markers (including but not limited to BRCA 1-2, ERCC 1-2-5, XRCC 1-2-3, RAD51 and 53BP1, PARP 1-2, P-histone H2AX and others) will be conducted. Statistical analysis will be performed to investigate the association between trial outcomes and polymorphisms of these genes.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Grignani, MD, Principal Investigator — Italian Sarcoma Group
Locations (3):
- Italy (3):
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Istituti Ortopedici Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - Istituto Nazionale Tumori - Unit of Medical Oncology, Milan

REFERENCES:
- [Result] Grignani G, D'Ambrosio L, Pignochino Y, Palmerini E, Zucchetti M, Boccone P, Aliberti S, Stacchiotti S, Bertulli R, Piana R, Miano S, Tolomeo F, Chiabotto G, Sangiolo D, Pisacane A, Dei Tos AP, Novara L, Bartolini A, Marchesi E, D'Incalci M, Bardelli A, Picci P, Ferrari S, Aglietta M. Trabectedin and olaparib in patients with advanced and non-resectable bone and soft-tissue sarcomas (TOMAS): an open-label, phase 1b study from the Italian Sarcoma Group. Lancet Oncol. 2018 Oct;19(10):1360-1371. doi: 10.1016/S1470-2045(18)30438-8. Epub 2018 Sep 11. PMID 30217671
- [Derived] Vyse S, Thway K, Huang PH, Jones RL. Next-generation sequencing for the management of sarcomas with no known driver mutations. Curr Opin Oncol. 2021 Jul 1;33(4):315-322. doi: 10.1097/CCO.0000000000000741. PMID 33927108